CLINICAL TRIAL: NCT01731808
Title: Outpatient Nurse Managed Counseling Program for Patients With Diabetic Foot Ulceration: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zurich University of Applied Sciences (Other)
Collaborators: Balgrist University Hospital (Other); Kantonsspital Winterthur KSW (Other); Luzerner Kantonsspital (Other); Kantonsspital Frauenfeld (Other); Spital Zollikerberg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Lorenz Imhof, Prof. Dr., Zurich University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2010-0278/0
Record Dates: First submitted 2012-10-18; First posted 2012-11-22 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Diabetic Foot Ulcer
Keywords: Nursing counseling; diabetic foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care (No Intervention): All participants received three specially-developed brochures with information regarding the diabetic foot condition. The brochures contained explanations to a) the cause and warning signs of diabetic foot ulcers, b) the precautions patients can take in their daily life, and c) helpful foot gymnastics to be practiced at home. The participants who were randomized in the control group received standard care. Standard care consisted of either physician-prescribed inpatient or outpatient wound care.
- Nursing counseling (Experimental)
  Interventions: Behavioral: Nursing counseling

INTERVENTIONS:
Behavioral: Nursing counseling — The participants who were randomized in the intervention group received outpatient physician-prescribed wound care. Additionally, they received standardized education regarding diabetic foot care. The nurse-led outpatient intervention started a few days after randomization and went on for five weeks. The study nurses conducting the interventions were wound care nurses and trained in foot examination, foot care, education, and counseling. During a period of five weeks, the participants were provided with weekly, one-hour education, skill training, and counseling sessions on foot care. Each participant received a foot care kit with essential foot care material and a foot care diary.
  Arms: Nursing counseling

SUMMARY:
The purpose of the study is to evaluate the feasibility and effectiveness of a physician directed nurse managed earlier outpatient counselling intervention for patients with diabetic foot ulceration.

For the purpose effectiveness is defined in two ways.1) as a reduction in hospital readmissions for complication for foot ulcers such as amputation or increased severity of the ulcer and 2) reduction in amputations, readmission rates. Selected covariates (self-efficacy,self-management, social support and depression) will be included to estimate predictors for readmission and amputation.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is associates with numerous complications. One of these is decreased peripheral circulation impaired sensation leading to the development of foot ulcers that lead to amputations of toes, feet and limbs. These complications not only have devastating effects on the individual in terms of loss of functionality but also impact the patient's ability to carry out and enjoy occupational, recreational and family functioning activities. Furthermore, foot ulcers and associated problems often lead to prolonged hospitalization and loss of productivity. All of these have personal as well as societal economical implications.

Currently, the standard of care includes admissions to the hospital lasting up to six weeks for medical observations and treatment of food ulcers.

The nursing responsibilities include daily or more frequent wound care as well as education counselling and skill building for diabetes self-management; therefore, an alternative to current practices must be considered. Such an alternative strategy has the potential benefit for the patient as well as the societal benefit of economic savings should such an outpatient nurse managed intervention be as or more effective as current practice. This type of service would allow the patients to remain in their home for care with probably a reduced risk for nosocomial infections.

This pilot randomized clinical trial (RCT) aims to evaluate the feasibility of an additional patient education program to current management of foot care in patients with DM. We plan to determine whether foot ulcer care in hospital under medical and nursing management can be improved by early discharge of the Intervention group (IG) to the well established outpatient wound care combined with an additional new outpatient nurse managed counselling program.

Expected results:

This study aims to test an alternative to current standard of care for patients with foot ulcers. A RCT is the preferred method to establish efficacy for this alternative nurse managed intervention; and if found to be effective, the current study will also allow an evaluation of the cost effectiveness of this intervention and the potential economic reduction in cost to the health care system.

Also, patients in the hospital are in danger of acquiring nosocomial infections, are subject to medical and nursing errors and are potentially accident prone; all of this together with a general preference for being able to live at home as compared to the hospital, together with the cost savings mentioned above could have a considerable impact on patient's quality of life, satisfaction with care, improvement in food ulcer and amputation outcomes.

Significance:

The potential implications are major in terms of quality of life, reduction in morbidity in disability days, and cost savings. It is anticipated that this intervention is at least as effective as hospital stay, and being surrounded by their own loved ones without the threats that a hospital setting presents. The findings will be important to consider whether clinical practice can be changed to benefit patients. If the study results show that the subjects in the IG have better skills in monitoring and treating their diabetic foot ulcerations and eventually avoid developing further complications the intervention can be applied to future patients.

ELIGIBILITY:
Inclusion Criteria:

* patients age 18 or older with
* current treatment for ulceration and/or amputation of a lower limb
* stable wound healing
* no signs of wound infection
* stable diabetes
* manageable pain

Exclusion Criteria:

* patients with cognitive impairment and psychiatric diseases
* patients living in dependent living facilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
feasibility of an intensive nurse led education program | The outcome measures will be assessed after all recruited participants have completed the five week education program - at the latest two years after study start.
  Recruitment procedures feasible yes/no; Randomization procedure feasible yes/no; Timeframe of the five week educational program feasible yes/no; Intervention material suitable yes/no

CONTACTS AND LOCATIONS:
Locations (5):
- Switzerland (5):
  - Kantonsspital Frauenfeld, Frauenfeld
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital Winterthur, Winterthur
  - Spital Zollikerberg, Zollikerberg
  - Uniklinik Balgrist, Zurich